CLINICAL TRIAL: NCT01224938
Title: Development and Validation of a Sputum Biomarker mRNA Panel for the Diagnostic Work-up of Asthma 1.
Acronym: BioSput-Air
Status: Completed | Type: Observational
Sponsor: Universitaire Ziekenhuizen KU Leuven (Other)
Responsible Party: Principal Investigator, Dominque Bullens, prof. dr., Universitaire Ziekenhuizen KU Leuven
Other Study IDs: Biomarker sputum airway study1
Record Dates: First submitted 2010-10-18; First posted 2010-10-20 (Estimated); Last update posted 2018-07-16 (Actual); Status verified 2018-07

CONDITIONS: Asthma Patients; Healthy Subjects

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples Without DNA — lysed sputum cells
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- Asthma patients: Asthmatics of all classes of severity will be included.
- Healthy control population: A healthy control population will be included to compare with the asthmatics.

SUMMARY:
The main objectives of the study are

1. to study the different T cell subtypes (Th1, Th2, Th17 and Treg) in the lower airways of healthy subjects and clinically different asthma patients, based on a non-invasive procedure of sputum induction. Patients will be different in function of age, in relation to the trigger (eg aspirin, without or with association with polyposis), without or with underlying atopic sensitization or different in the type of underlying inflammation (eosinophilic vs neutrophilic). This T cell pattern will become the basis of molecular phenotyping in the patients.
2. to study the usefulness of asthma molecular phenotyping (by following the balance between the inflammatory markers on the one hand and the regulatory markers on the other hand) in asthma guidance (longitudinally).

The final goal of this project is then to develop a sputum non-invasive biomarker array that can be used to distinguish the different inflammatory asthma phenotypes and that can predict steroid resistance and/or sensitivity to other anti-inflammatory medication, using a non-invasive technique that can be used also at young age and repetitively.

ELIGIBILITY:
Inclusion Criteria:

* asthma diagnosis

Exclusion Criteria:

* viral/bacterial/fungal infection with fever (<1 month )
* other airway diseases (CF, ciliar dyskinesia, bronchiectasis)
* asthma exacerbation (<3 months)

Ages: 6 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: 330 asthmatics (300 adults, 30 children) will be recruited from the outpatient clinic of the university hospital of Leuven. 115 healthy subjects (100 adults, 15 children) will be recruited among students and co-workers from the KULeuven and UZ Leuven.
Sampling Method: Probability Sample
Enrollment: 395 (Actual)
Dates: Start 2010-10; Primary Completion 2012-03 (Actual); Study Completion 2013-09 (Actual)

PRIMARY OUTCOMES:
sputum cytokine mRNA | one year

SECONDARY OUTCOMES:
lung function parameters | one year
asthma symptom scores | one year
non-invasive measurements of airway inflammation | one year

CONTACTS AND LOCATIONS:
Overall Officials: Dominique MA Bullens, MD, PhD, Principal Investigator — Lab of clinical immunology, O&N I Herestraat 49 - bus 811, 3000 Leuven, België; Sven F Seys, MSc, Study Director — Lab of clinical immunology, O&N I Herestraat 49 - bus 811, 3000 Leuven, België
Locations (1):
- University Hospital of Leuven, Leuven, Vlaams-Brabant, Belgium

REFERENCES:
- [Background] Bullens DM, Decraene A, Dilissen E, Meyts I, De Boeck K, Dupont LJ, Ceuppens JL. Type III IFN-lambda mRNA expression in sputum of adult and school-aged asthmatics. Clin Exp Allergy. 2008 Sep;38(9):1459-67. doi: 10.1111/j.1365-2222.2008.03045.x. Epub 2008 Jun 28. PMID 18564328
- [Background] Bullens DM. Measuring T cell cytokines in allergic upper and lower airway inflammation: can we move to the clinic? Inflamm Allergy Drug Targets. 2007 Jun;6(2):81-90. doi: 10.2174/187152807780832210. PMID 17692031
- [Background] Bullens DM, Truyen E, Coteur L, Dilissen E, Hellings PW, Dupont LJ, Ceuppens JL. IL-17 mRNA in sputum of asthmatic patients: linking T cell driven inflammation and granulocytic influx? Respir Res. 2006 Nov 3;7(1):135. doi: 10.1186/1465-9921-7-135. PMID 17083726
- [Background] Truyen E, Coteur L, Dilissen E, Overbergh L, Dupont LJ, Ceuppens JL, Bullens DM. Evaluation of airway inflammation by quantitative Th1/Th2 cytokine mRNA measurement in sputum of asthma patients. Thorax. 2006 Mar;61(3):202-8. doi: 10.1136/thx.2005.052399. Epub 2006 Jan 31. PMID 16449261
- [Result] Seys SF, Scheers H, Van den Brande P, Marijsse G, Dilissen E, Van Den Bergh A, Goeminne PC, Hellings PW, Ceuppens JL, Dupont LJ, Bullens DM. Cluster analysis of sputum cytokine-high profiles reveals diversity in T(h)2-high asthma patients. Respir Res. 2017 Feb 23;18(1):39. doi: 10.1186/s12931-017-0524-y. PMID 28231834
- [Derived] Goossens J, Jonckheere AC, De Boodt S, Dilissen E, Marain N, Decaesteker T, Cortes A, Vanoirbeek JA, Seys SF, Dupont L, Bullens DMA. Sputum Transcriptomic Analysis and Clustering Reveals Insight Into Asthma Heterogeneity. Lung. 2025 Aug 20;203(1):89. doi: 10.1007/s00408-025-00843-1. PMID 40830242